CLINICAL TRIAL: NCT05731908
Title: Pharmacokinetics, Safety, and Tolerability of BI 690517 in Subjects With Mild and Moderate Liver Impairment (Child-Pugh Classification A and B) as Compared to Healthy Subjects
Brief Title: A Study to Test How BI 690517 is Taken up in the Body of People With and Without Liver Problems
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: IQVIA global CRO (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1378-0016
Record Dates: First submitted 2023-02-08; First posted 2023-02-16 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Liver Diseases; Healthy
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BI 690517 mild hepatic impairment (Child-Pugh A) (Experimental)
  Interventions: Drug: BI 690517
- BI 690517 normal hepatic function (Experimental): control group
  Interventions: Drug: BI 690517
- BI 690517 moderate hepatic impairment (Child-Pugh B) (Experimental)
  Interventions: Drug: BI 690517

INTERVENTIONS:
Drug: BI 690517 — BI 690517
  Other Names: Vicadrostat

SUMMARY:
The main objective of this trial is to assess the effect of mild and moderate hepatic impairment (Child-Pugh classification A and B) on the pharmacokinetics, safety, and tolerability of BI 690517 in comparison with a control group with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged at least 18 years at screening
* Body mass index of 18.5 to 36.0 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
* Women of childbearing potential1 and men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.

Inclusion criteria applying only to participants with impaired hepatic function:

* Hepatic impairment classified as Child-Pugh A (score 5-6 points) or Child-Pugh B (score 7-9 points)
* Absence of clinically significant abnormalities, as based on a complete medical history including a full physical examination, vital signs (Blood pressure, Pulse rate), 12-lead Electric Cardiogram, and clinical laboratory tests at both screening and admission to trial site, with the exception of findings that in the opinion of the investigator are consistent with the participant's hepatic impairment.
* Medication and/or treatment regimens must have been stable (i.e., no dose adjustments) for at least 4 weeks prior to the screening period and should be kept stable until study completion. Fluctuating treatment regimens may be considered for inclusion on a case-by-case basis if the underlying disease is under control in the opinion of the investigator and must be agreed to by both the investigator and the sponsor's medical monitor.

Inclusion criteria applying only to healthy participants with normal hepatic function:

* Healthy subjects according to the following criteria: the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests.
* Individually matched to participants with hepatic impairment according to sex, age, and weight

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurements of blood pressure and pulse rate out of range considered clinically significant by the investigator
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, except for laboratory values outside the reference range due to underlying disease
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except cholecystectomy, appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Relevant chronic or acute infections
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 4 days
Maximum measured concentration of the analyte in plasma (Cmax) | Up to 4 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to 4 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Omega Research Orlando, LLC, Orlando, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com